CLINICAL TRIAL: NCT06613646
Title: The Importance of Pectoralis Minor Syndrome in Hemiplegic Shoulder Pain: A Prospective, Interventional Study
Brief Title: The Importance of Pectoralis Minor Syndrome in Hemiplegic Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Burak Ugur Cetin, Medical Doctor, Istanbul University - Cerrahpasa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IstanbulUC-BCetin-01
Record Dates: First submitted 2024-09-12; First posted 2024-09-26 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Hemiplegic Shoulder Pain; Pectoralis Minor Syndrome
Keywords: Pectoralis Minor Syndrome; Ultrasound Guided Injections; Hemiplegia; Hemiplegic Shoulder Pain
MeSH Terms: conditions — Hemiplegia | interventions — Lidocaine; Pharmaceutical Preparations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): Patients presenting to the outpatient clinic with shoulder pain on the hemiplegic side will first undergo a diagnostic subacromial bursa injection, followed by a pectoralis minor muscle block.
  Interventions: Procedure: Ultrasound-guided injection of the subacromial bursa and pectoralis minor; Drug: Lidocaine (drug)

INTERVENTIONS:
Procedure: Ultrasound-guided injection of the subacromial bursa and pectoralis minor — Patients will first receive an ultrasound-guided injection of the subacromial bursa. After the subacromial bursa injection, patients will be monitored for 1 hour, after which the level of relief in their complaints will be assessed using the Numeric Rating Scale (NRS), and passive range of motion will be measured.
  Following the subacromial bursa injection, patients will receive an ultrasound-guided injection of the pectoralis minor muscle. After the pectoralis minor muscle injection, patients will again be monitored for 1 hour, after which the level of relief in their complaints will be assessed using the NRS, and passive range of motion will be measured.
Drug: Lidocaine (drug) — 5 mL of 2% lidocaine will be used as a local anesthetic for the subacromial bursa injection, and 4 mL of 2% lidocaine will be used for the pectoralis minor muscle injection.

SUMMARY:
Hemiplegic shoulder pain, common in stroke patients, often arises from muscle weakness, imbalance, or joint and nerve issues. Previous case reports in literature suggest that pectoralis minor syndrome may play a significant role in this pain. In current study, the investigators aimed to evaluate the role of the pectoralis minor muscle in patients with hemiplegic shoulder pain and to reveal the contribution of pectoralis minor syndrome to hemiplegic shoulder pain. Additionally, this study may provide fundamental information to improve clinical practice in determining rehabilitation and treatment strategies, contribute to the development of new approaches in managing hemiplegic shoulder pain, and assist in optimizing rehabilitation programs.

DETAILED DESCRIPTION:
Hemiplegic shoulder pain is a common complication following a stroke, with a prevalence ranging from 22% to 47%, typically occurring two to three months post-stroke. This pain can lead to withdrawal from rehabilitation programs, longer hospital stays, reduced joint mobility, and impaired quality of life. Various factors contribute to its development, including decreased muscle tone, shoulder subluxation, increased muscle tone, impingement syndrome, frozen shoulder, brachial plexus injury, and thalamic syndrome. Among these, subacromial/subdeltoid bursitis is the most frequently reported cause of pain, and significant pain relief following local anesthetic injections into the subacromial/subdeltoid bursa is diagnostic of subacromial impingement syndrome.

Treatment goals for hemiplegic shoulder pain include pain reduction, restoring shoulder mobility, improving functional activities, and preventing degenerative changes. Treatment options range from conservative methods like shoulder slings, range-of-motion exercises, pain relievers, physical therapy, and various injection therapies, to surgical interventions for cases unresponsive to conservative measures.

Pectoralis minor syndrome, associated with hemiplegic shoulder pain, can occur in stroke patients. The pectoralis minor muscle plays a crucial role in shoulder stability and movement. Compression or irritation of neurovascular structures in the retropectoral space by this muscle leads to pectoralis minor syndrome, often diagnosed through clinical evaluation rather than specific radiological or electrophysiological tests. Ultrasound-guided pectoralis minor muscle blocks have become significant in both diagnosis and treatment, demonstrating marked pain reduction in affected patients. Research on pectoralis minor syndrome aims to enhance understanding of its causes, effects, and treatment strategies, contributing to the development of more effective and specific approaches for managing hemiplegic shoulder pain.

ELIGIBILITY:
Inclusion Criteria:

* Development of spastic hemiplegia due to stroke
* Presence of shoulder pain on the hemiplegic side

Exclusion Criteria:

* Lack of medical stability
* Inability to communicate verbally
* History of severe sensitivity to lidocaine injections
* Surgical history related to the hemiplegic shoulder
* Presence of a prosthesis in the hemiplegic shoulder
* Malignancy in the hemiplegic shoulder
* Severe psychiatric illness
* History of injections to the hemiplegic shoulder within the last 6 months
* Pregnancy
* History of inflammatory rheumatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
Pain Relief | Baseline, one hour after subacromial bursa injection, one hour after pectoralis minor injection, one week, and one month
  Pain will be assessed using the Numerical Rating Scale (NRS), which ranges from 0 (no pain) to 10 (worst pain imaginable), at rest, during movement, at night, and overall, both before and after injections into the subacromial bursa and the pectoralis minor muscle. Higher scores indicate worse pain outcomes.
Passive Range of Motion of Shoulder | Baseline, one hour after subacromial bursa injection, one hour after pectoralis minor injection, one week, and one month
  Passive shoulder flexion, abduction, and external rotation will be measured with a goniometer. Flexion and abduction will be measured from 0° (no range of motion) to 180° (full range of motion), while external rotation will be measured from 0° to 90°. Higher scores indicate better outcomes in terms of range of motion.

SECONDARY OUTCOMES:
Modified Ashworth Scale | Baseline
  Spasticity in upper extremity muscles will be assessed using the Modified Ashworth Scale (MAS), which ranges from 0 to 4. A score of 0 indicates no increase in muscle tone, while a score of 4 indicates the affected part is rigid in flexion or extension. Higher scores on the MAS indicate worse spasticity outcomes.
Brunnstrom Stages of Recovery for Upper Extremity Motor Function and Hand Function | Baseline
  Upper extremity motor function and hand function will be assessed using the Brunnstrom Stages of Recovery. This scale ranges from Stage 1 (flaccidity, no voluntary movement) to Stage 6 (normal motor function). For both upper extremity motor function and hand function, higher scores indicate better recovery and motor outcomes.
Functional Ambulation Scale | Baseline
  Ambulation will be assessed using the Functional Ambulation Scale, which ranges from 0 to 5. A score of 0 indicates the inability to walk or requiring maximal assistance, while a score of 5 indicates independent ambulation on all surfaces without assistance. Higher scores indicate better ambulation outcomes.
Subluxation in the glenohumeral joint | Baseline
  It will be assessed by placing the ultrasound probe along the long axis of the humerus over the lateral edge of the acromion. The distance is defined as the relative lateral distance between the lateral edge of the acromion and the nearest edge of the superior part of the greater tuberosity of the humerus. A difference greater than 0.4 cm indicates the presence of subluxation.
Overall Improvement | One hour after subacromial bursa injection, one hour after pectoralis minor injection, one week, one month
  Overall improvement will be assessed as a self-reported percentage, ranging from 0% (no improvement) to 100% (complete improvement). Higher percentages indicate better outcomes, with 100% representing full recovery as perceived by the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University - Cerrahpasa (IUC), Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Neer CS 2nd. Impingement lesions. Clin Orthop Relat Res. 1983 Mar;(173):70-7. No abstract available. PMID 6825348
- [Result] Aktas I, Kaya E, Akpinar P, Atici A, Unlu Ozkan F, Palamar D, Akgun K. Spasticity-induced Pectoralis minor syndrome: a case-report. Top Stroke Rehabil. 2020 May;27(4):316-319. doi: 10.1080/10749357.2019.1691807. Epub 2019 Nov 27. PMID 31774031
- [Result] Lin PH. Sonographic findings of painful hemiplegic shoulder after stroke. J Chin Med Assoc. 2018 Jul;81(7):657-661. doi: 10.1016/j.jcma.2017.07.018. Epub 2017 Dec 6. PMID 29217360
- [Result] Sanders RJ, Annest SJ. Thoracic outlet and pectoralis minor syndromes. Semin Vasc Surg. 2014 Jun;27(2):86-117. doi: 10.1053/j.semvascsurg.2015.02.001. Epub 2015 Feb 18. PMID 25868762
- [Result] Lee KW, Choi YJ, Lee HJ, Gil YC, Kim HJ, Tansatit T, Hu KS. Classification of unusual insertion of the pectoralis minor muscle. Surg Radiol Anat. 2018 Dec;40(12):1357-1361. doi: 10.1007/s00276-018-2107-0. Epub 2018 Oct 10. PMID 30306210
- [Result] Murie-Fernandez M, Carmona Iragui M, Gnanakumar V, Meyer M, Foley N, Teasell R. [Painful hemiplegic shoulder in stroke patients: causes and management]. Neurologia. 2012 May;27(4):234-44. doi: 10.1016/j.nrl.2011.02.010. Epub 2011 Apr 22. Spanish. PMID 21514698
- [Result] Adey-Wakeling Z, Arima H, Crotty M, Leyden J, Kleinig T, Anderson CS, Newbury J; SEARCH Study Collaborative. Incidence and associations of hemiplegic shoulder pain poststroke: prospective population-based study. Arch Phys Med Rehabil. 2015 Feb;96(2):241-247.e1. doi: 10.1016/j.apmr.2014.09.007. Epub 2014 Sep 28. PMID 25264111
- [Result] Lindgren I, Jonsson AC, Norrving B, Lindgren A. Shoulder pain after stroke: a prospective population-based study. Stroke. 2007 Feb;38(2):343-8. doi: 10.1161/01.STR.0000254598.16739.4e. Epub 2006 Dec 21. PMID 17185637
- [Result] Griffin JW. Hemiplegic shoulder pain. Phys Ther. 1986 Dec;66(12):1884-93. doi: 10.1093/ptj/66.12.1884. PMID 2431421
- [Result] Bender L, McKenna K. Hemiplegic shoulder pain: defining the problem and its management. Disabil Rehabil. 2001 Nov 10;23(16):698-705. doi: 10.1080/09638280110062149. PMID 11732559